CLINICAL TRIAL: NCT04599621
Title: Immunological Features of Unstable Angina Pectoris in Comorbidity With Anxiety-depressive Syndrome
Brief Title: Unstable Angina Pectoris in Comorbidity With Anxiety-depressive Syndrome
Status: Recruiting | Type: Observational
Sponsor: Samarkand State Medical Institute (Other)
Responsible Party: Sponsor
Other Study IDs: DGU20191075
Record Dates: First submitted 2020-10-06; First posted 2020-10-23 (Actual); Last update posted 2020-10-23 (Actual); Status verified 2020-04

CONDITIONS: Coronary Heart Disease
Keywords: unstable angina pectoris; uric acid; cytokine imbalance
MeSH Terms: conditions — Coronary Disease; Angina, Unstable

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — All study participants had blood in the morning on fasting after 8-12 hours of fasting from the cubital vein. Determination of the level of cytokines TNF-α, IL-1β, IL-4 and IL-10 in blood serum by enzyme-linked immunosorbent assay (ELISA).
  Sample preparation: before testing, 1 part of the plasma is diluted 30-50 times with Tris buffer, depending on the test system and the kit manufacturer's instructions.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (1):
- patients with unstable angina: This group included patients with frequent anginal attacks, with a burdened history and comorbid conditions.
  Interventions: Diagnostic Test: Collection of blood samples to determine the level of certain cytokines (TNF-α, IL-1β, IL-4 and IL-10),Collection of blood samples to determine the level of uric acid

INTERVENTIONS:
Diagnostic Test: Collection of blood samples to determine the level of certain cytokines (TNF-α, IL-1β, IL-4 and IL-10),Collection of blood samples to determine the level of uric acid — Collection of blood samples to determine the level of certain cytokines (TNF-α, IL-1β, IL-4 and IL-10) All study participants had blood in the morning on fasting after 8-12 hours of fasting from the cubital vein. Determination of the level of cytokines TNF-α, IL-1β, IL-4 and IL-10 in blood serum by enzyme-linked immunosorbent assay (ELISA). All participants in the study had blood drawn in the morning on fasting after 8-12 hours of fasting from the cubital vein. The level of uric acid was determined on the CYAN Start apparatus using a unified method.

SUMMARY:
Introduction:

Today it is necessary to emphasize that coronary heart disease is often associated with anxiety disorders. Research over the years has shown several and sometimes surprising links between coronary heart disease and mental illness, and has even suggested that both of these phenomena may actually cause each other. However, the exact nature of these links has not yet been clearly established.

Methods: The study included 202 patients with coronary artery disease, of whom 42 patients were with stable angina pectoris, they participated as a control group, and 160 patients with unstable angina pectoris, who made up the main group.

Among them there are 102 women and 100 men between the ages of 30 and 88. The average age was 63.75 ± 11.37 years.

All study participants had blood in the morning on fasting after 8-12 hours of fasting from the cubital vein. Determination of the level of cytokines TNF-α, IL-1β, IL-4 and IL-10 in blood serum by enzyme-linked immunosorbent assay (ELISA).

All participants in the study had blood drawn in the morning on fasting after 8-12 hours of fasting from the cubital vein. The level of uric acid was determined on the CYAN Start apparatus using a unified method.

When examining patients with unstable angina pectoris were used: hospital anxiety and depression scale [Kozlova S.N. 2013]. And also the Spielberger-Khanin scale [Psychiatry - Hoffman A.G. 2010], developed by Spielberger Ch.D. and adapted by Yu.L. Khanin. to assess cognitive functions [Psychiatry - Gofman A.G. 2010].

DETAILED DESCRIPTION:
All study participants had blood in the morning on fasting after 8-12 hours of fasting from the cubital vein. Determination of the level of cytokines TNF-α, IL-1β, IL-4 and IL-10 (pg/ml) in blood serum by enzyme-linked immunosorbent assay (ELISA).

Sample preparation: before testing, 1 part of the plasma is diluted 30-50 times with Tris buffer, depending on the test system and the kit manufacturer's instructions.

Definition progress:

1. preparation of microtiter strips;
2. add the material diluted with buffer to the well of the microtiter strip and incubate for 1 hour at room temperature;
3. washing;
4. add immunoconjugates to the well of the microtiter strip and incubate for 1 hour at room temperature;
5. washing;
6. add the o-phenyldiamine / H2O2 substrate solution;
7. after exactly 3 minutes of hydrochloric acid (1 mol / l);
8. reading the results on an ELISA analyzer after 10-120 minutes. 2.4. Collection of blood samples to determine the level of uric acid All participants in the study had blood drawn in the morning on fasting after 8-12 hours of fasting from the cubital vein. The level of uric acid was determined on the CYAN Start apparatus using a unified method.

2.5. Method for determining anxiety-depressive syndrome. When examining patients with unstable angina pectoris were used: Hospital scale [Kozlova S.N. 2013]. And also the Spielberger-Khanin scale [Psychiatry - Hoffman A.G. 2010], developed by Spielberger Ch.D. and adapted by Yu.L. Khanin. to assess cognitive functions [Psychiatry - Gofman A.G. 2010].

Description of the hospital scale This questionnaire is intended for self-completion by the patient [Kozlova S.N. 2013]. The questionnaire consists of 14 statements, "serving" 2 subscales: the subscale "alarm" marked in red, consists of odd items - 1, 3, 5, 7, 9, 11, 13 and the subscale "depression" marked in blue consists of even items - 2, 4, 6, 8, 10, 12, 14.

Each statement corresponds to 4 answer options, reflecting gradations of the severity of the sign and coded according to the increase in the severity of the symptom from 0 (no) to 3 (maximum severity). The final scores for the two subscales are obtained by summing the numerical values of the answers. When interpreting the results, the total indicator for each subscale is taken into account, while there are 3 areas of its values:

* 0-7 - normal (no reliably pronounced symptoms of anxiety and depression);
* 8-10 - subclinical anxiety and / or depression;
* 11 and above - clinically significant anxiety and / or depression. The filling of the scale was carried out by patients under standard conditions, after a short instruction for filling, within a clear time frame.

Description of the Spielberger-Hanin scale The Spielberger Anxiety Scale is an informative way to self-assess the level of anxiety at a given moment (reactive anxiety as a state) and personal anxiety (as a stable characteristic of a person). Developed by Ch.D.Spielberger and adapted by Yu.L. Khanin [Psychiatry - Gofman A.G. 2010].

This scale consists of two subscales: judgments from 1 to 20 determine the presence of situational anxiety, judgments from 21 to 40 determine the presence of personal anxiety.

When analyzing the results of self-assessment, it should be borne in mind that the overall final indicator for each of the subscales can range from 20 to 80 points. Moreover, the higher the final indicator, the higher the level of anxiety (situational or personal).

When interpreting indicators, you can use the following rough estimates of anxiety:

* up to 40 points - low,
* 41 - 54 points - moderate;
* 55 and more - high. 2.6. Treatment All patients with unstable angina pectoris offer conventional therapy, which includes intravenous infusion of nitrates for 12-24 hours, followed by prolonged nitrates, beta-blockers, ACE inhibitors or sartans, antiplatelet agents, anticoagulants, clopidogrel, statins. Patients have elevated levels of uric acid according to the traditional immedia Febuxostat (not a purine blocker of xanthine oxide, manufactured by Berlin Chemie, Germany) at a dose of 0.04-0.08 g / day per day. Patients who had anxiety-depressive syndrome Divase syndrome (antibodies to the brain-specific protein S-100, manufacturer MATERIA MEDICA HOLDING, LLC (Russia)) in a fixed dose of 0.6 mg / day, which has a neurotropic and antioxidant effect.

ELIGIBILITY:
Inclusion Criteria:

* the presence of an established diagnosis in patients with coronary artery disease
* unstable angina pectoris (NS). When making a diagnosis, the recommendations of ESH / ESC (2015) and RCO / WHO (2014) were used.
* stable exertional angina (SSN) I-III FC. When making the diagnosis, the IHD classification was used, adopted at the IV Congress of Cardiologists of the Republic of Uzbekistan (2000), as well as in accordance with the recommendations of ESH / ESC (2019) and RCO / WHO (2017)

Exclusion Criteria:

* The patient's refusal to participate in the study;
* Pregnancy and lactation;
* Severe and unstable condition of the patient, making it difficult to conduct a questionnaire (for ethical reasons);
* Acute violation of cerebral circulation;
* History of acute or chronic psychosis;
* The presence of concomitant acute diseases or chronic diseases in the acute stage.

Throughout the study, all patients were assigned the right to voluntarily withdraw from the study at their own request, notifying the researcher in writing or orally.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: When collecting anamnesis in patients with unstable angina pectoris, the presence of ischemic heart disease (previous MI, exertional or rest angina pectoris), the presence of risk factors for coronary artery disease and myocardial infarction (atherosclerosis of other vascular areas, hypertension, smoking, diabetes mellitus, obesity) was determined. When questioning the patient, attention was paid to the period preceding the development of myocardial infarction, as well as the factors that provoked the development of this disease (excessive physical activity, infections, psychoemotional stress), as well as information on the early manifestation of CVD in the closest relatives.
Sampling Method: Non-Probability Sample
Enrollment: 3 (Estimated)
Dates: Start 2018-11-05 (Actual); Primary Completion 2025-12-25 (Estimated); Study Completion 2027-12-28 (Estimated)

PRIMARY OUTCOMES:
cytokine research | 2019-2027
  Determination of the level of cytokines TNF-α, IL-1β, IL-4 and IL-10 in blood serum was performed by enzyme-linked immunosorbent assay (ELISA). The principle of operation of the test system for the determination of cytokines is based on the "sandwich" method of solid-phase immune enzyme immunoassay using horseradish peroxidase as an indicator enzyme. Stop the reaction by adding 50 μl of 1N sulfuric acid solution. The quantitative assessment of the results is carried out by the method of constructing a calibration curve or using a commercial computer program "Microplate manager", reflecting the dependence of optical density on concentration for a standard antigen and allowing comparison of the test samples with it. The sensitivity of the method is 5-30 pg / ml.
hospital scale | 2019-2027
  The questionnaire consists of 14 questions, 2 subscales. 0-7 - normal, 8-10 - subclinical anxiety or depression; 11 and above - clinically significant anxiety or depression.
Spielberger-Khanin Anxiety Scale | 2019-2027
  The scale consists of 2 subscales: judgments from 1 to 20 determine situational anxiety, judgments from 21 to 40 determine the presence of personal anxiety. The results for each subscale can be from 20 to 80 points. up to 40 points - low, 41 - 54 points - moderate; 55 and more - high.

SECONDARY OUTCOMES:
etermination of uric acid level | 2019-2027
  Method: Enzymatic Uricase Colorimetric Method Analyzer: Cobas 6000 Measurement units: μmol / l Material for research: venous blood serum
  Training:
  Take on an empty stomach (after sleep and 8-12 hours of fasting). It is permissible to drink only pure non-carbonated water (up to 200 ml) (with the exception of glucose analysis).
  Do not eat spicy, fatty, fried foods for 1-2 days before analysis. Eliminate physical and emotional stress 1 day before the analysis. Do not smoke for at least 1 hour before analysis. It is not recommended to take it after radiography, physiotherapy procedures and instrumental examinations.
  For several days before the study, you must adhere to a low-purine diet, avoid drinking alcohol or warn about the use when taking a test.

CONTACTS AND LOCATIONS:
Locations (1):
- Zarina, Samarkand, Uzbekistan

IPD SHARING:
Plan to Share IPD: Undecided
For the first time in the region of Uzbekistan, the mechanisms of interconnection of biopsychosocial risk factors affecting the progression of coronary heart disease, taking into account the level of uric acid in the blood and cytokine imbalance, will be studied. Indicators of cytokine status will be identified that affect the progression of coronary heart disease depending on the level of uric acid in the blood